CLINICAL TRIAL: NCT04238585
Title: Intervening to Promote Healthy Weight From Gestation to Age 2, Particularly Among Disproportionately Burdened Populations
Brief Title: BabyQ's: Randomized Controlled Trial of Health Messaging in Pregnancy and Infancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Woo Baidal, Assistant Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: AAAS0859
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Pregnancy Related; Infant Development
Keywords: Sugar-sweetened beverages; Early life nutrition; First 1000 Days

STUDY DESIGN:
Intervention Model Description: Families who present for a routine WIC visit will be referred for study staff recruitment if they meet either of the following criteria: 1) pregnant woman or 2) parent of child <24 months enrolled in WIC.
Who Masked: Participant, Investigator
Masking Description: Research staff performing data collection will be blinded to the intervention arm of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Negative message frames (Active Comparator): Participants will receive messages framed in a negative manner to avoid sugar-sweetened beverages
  Interventions: Behavioral: Mobile messaging
- Sugar content information messages (Active Comparator): Participants will receive messages framed in a positive manner to promote healthy beverage consumption
  Interventions: Behavioral: Mobile messaging
- Attention Control-Infant Safety (Placebo Comparator): Participants will receive messages with infant safety education materials-attention control group
  Interventions: Behavioral: Mobile messaging

INTERVENTIONS:
Behavioral: Mobile messaging — Mobile health messages

SUMMARY:
This randomized controlled intervention evaluates the effect of a mobile health behavioral intervention to test messages to reduce sugar-sweetened beverage intake during pregnancy and infancy.

The study team will perform a prospective, longitudinal, interventional, randomized control trial by recruiting 300 WIC families during the first 1,000 days of life (pregnancy through infant age 2 months) at consecutive Women, Infants, and Children (WIC) visits to test two interventions compared to a control group. The study team will implement a mobile-based messaging intervention allocate participants to one of 3 arms for a 1 month period: 1) negative message frames, 2) positive message frames, and 3) attention control.

DETAILED DESCRIPTION:
Childhood obesity prevalence soared over the past four decades with a 10-fold increase globally from 1975-2015 and Healthy People 2020 has declared obesity a national health priority. Socioeconomic and racial/ethnic disparities in obesity exist and may be widening. These disparities are apparent by age 2 years with recent national data showing that Hispanic children continue to have highest obesity prevalence (15.6%) and on-Hispanic black children have 2-fold higher obesity prevalence (10.4%) compared to non-Hispanic white (5.2%) counterparts. The first 1,000 days describes the period from pregnancy through child age 2 years, and is increasingly recognized as a critical period for development of childhood obesity and its adverse consequences. Several risk factors are consistently associated with later childhood obesity during the first 1,000 days and are more prevalent among low socioeconomic groups and racial/ethnic minorities. These modifiable risk factors mediate the development of racial/ethnic disparities in later childhood obesity.

Sugar-sweetened beverage (SSB) consumption during the first 1,000 days is a risk factor for childhood overweight/obesity, and has been linked to dental caries, lower child cognition, and the adverse child health consequences. Recent evidence shows that maternal SSB consumption during pregnancy and infant SSB consumption in the first year of life are associated with childhood obesity later in life. Thus, interventions to curb SSB consumption and promote healthy beverage intake in urban, low-income Hispanic/Latino families must start early in life, yet few SSB-specific interventions have ventured to do so.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years or older or; legal caretakers of infants under 24 months enrolled in WIC
* Can respond to questions in English or Spanish
* Report use of a mobile device using iOS or Android
* Give permission to enroll in messaging system

Exclusion Criteria:

* Pregnant women with chronic medical conditions that may impact their nutrition behaviors
* Families whose eligible child has chronic conditions that interest with growth or feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Change in sugar-sweetened beverage (SSB) intake in kcals among adult participants | 1 month
  Determine change from baseline to follow-up in habitual daily caloric intake of SSBs using parent self report of beverage intake

SECONDARY OUTCOMES:
Change in sugar-sweetened beverage (SSB) intake in infants | 1 month
  Determine change from baseline to follow-up in parent-reported infant SSB intake using logistic regression to examine a categorical outcome (any infant SSB consumption v. none)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Woo Baidal, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No